CLINICAL TRIAL: NCT02562105
Title: In a Developing Country; What is the Fate of Hematologic Cancer Patients Requiring Mechanical Ventilation for More Than One Day? A Prospective Cohort Study
Brief Title: Prognosis of Hematological Cancer Patient Underwent Mechanical Ventillation
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Enas Aly Abd El motlb, Assistant professor, Mansoura University
Other Study IDs: 15.05.42
Record Dates: First submitted 2015-09-23; First posted 2015-09-29 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Hematological Malignancy; Acute Respiratory Failure; Mechanical Ventilation
Keywords: Intensive care unit; Hematological malignancy; Acute respiratory failure; Prognosis; Mechanical ventilation
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Mechanical ventilation: requiring mechanical ventilation at admission to ICU for one day or more during the study period
  Interventions: Procedure: Mechanical ventilation

INTERVENTIONS:
Procedure: Mechanical ventilation — requiring mechanical ventilation at admission to ICU for one day or more during the study period

SUMMARY:
This observational cohort aimed to re-evaluate the outcome of hematologic cancer patients admitted to the intensive care unit of Mansoura oncology center through a cohort study as regards their need for mechanical ventilation during two years.

DETAILED DESCRIPTION:
It has been believed for many years that the scene of cancer patients requiring mechanical ventilation is frustrating. The needed life support measures drain much of health resources and add a significant burden on the patient's family. Many factors have been responsible for the high mortality rates among hematologic cancer patients admitted to intensive care unit. Among of these factors, the invasive treatments that are frequently employed in today's intensive care unit. These procedures give chance for development of severe infection and multiple organ failure which are common events in immune-compromised patients (e.g. neutropenia) and in those exposed to chemotherapy. The most common form of organ failure in those patients is acute respiratory failure which is a major predictor of mortality in that population. The prognosis of such failure may vary depending on its causes and severity, co morbidity, associated acute organ failure and characters of the underlying malignancy. After the recent advances in the field of intensive care and shedding light on the benefits of the noninvasive ventilation in immune-compromised patients, the overall survival rate of cancer patients admitted to intensive care unit are improving.

ELIGIBILITY:
Inclusion Criteria:

* Critical ill hematological cancer patient
* Requiring mechanical ventilation

Exclusion Criteria:

* Patients with acute coronary syndrome.
* Patients with cancer remission more than 5 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hematological cancer patients admitted to ICU of oncology center, Mansoura University
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Survival | through study completion, an average of 30 days after admission to intensive care unit
  Continuing to live

SECONDARY OUTCOMES:
Sequential Organ Failure Assessment score | up to 24 hours after admission to the intensive care unit
  Sequential Organ Failure Assessment (SOFA) Score
Simplified Acute Physiology Score II | up to 24 hours after admission to the intensive care unit
  Simplified Acute Physiology Score (SAPS II)
Mode of mechanical ventilation | up to 24 hours after admission to the intensive care unit
  synchronised intermittent, pressure-controlled, volume-controlled, pressure support, continuous positive airway pressure, volume guarantee, adjusted pressure release ventilation, or adaptive proportional assist ventilation
lowest Pa02/FiO2 | up to 24 hours after admission to the intensive care unit
  PaO2 "arterial oxygen tension"/FiO2 "inspired fraction of oxygen" ratio
Reason for need of ventilatory support | up to 24 hours after admission to the intensive care unit
  Advanced malignancy, respiratory muscle weakness, respiratory failure, lung metastasis, coma, sepsis, multi-organs failure

OTHER OUTCOMES:
Associated comorbidities | up to 24 hours after admission to the intensive care unit
  Like as sepsis, acute respiratory distress syndorme, or leukopenia
Cancer status | up to 24 hours after admission to the intensive care unit
  Early or advanced stage

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Enas A Abd El motlb, MD, Principal Investigator — Mansoura University, College of Medicine
Locations (1):
- Mansoura Cancer Therapy Center, Al Mansurah, Dakahlia Governorate, Egypt